CLINICAL TRIAL: NCT04860479
Title: Evaluation of a Femoralis, n Femoralis and m Iliopsoas Tendon Sonoanatomy According to Age Groups in Children
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Collaborators: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hande Gurbuz, Medical Doctor, Associate Professor, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Anatomic Abnormality; Anatomy; Pediatrics; Anatomic Landmarks; Anthropometry
Keywords: sonoanatomy; pediatrics; inguinal region; variation; anatomy; PENG; femoral nerve; regional anesthesia; femoral artery
MeSH Terms: conditions — Congenital Abnormalities | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Infants: 28 days - 12 month: inguinal sonoanatomy
  Interventions: Device: ultrasound
- small children: 13 months - 36 months: inguinal sonoanatomy
  Interventions: Device: ultrasound
- preschool age: 37 months - 72 months: inguinal sonoanatomy
  Interventions: Device: ultrasound
- school age: 73 months - 9 years: inguinal sonoanatomy
  Interventions: Device: ultrasound
- Preadolescant: >9 years - 12 years: inguinal sonoanatomy
  Interventions: Device: ultrasound
- Adolescants: >12 years - 18 years: inguinal sonoanatomy
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — ultrasonography to inguinal region

SUMMARY:
This study aims to examine the sonoanatomy of the inguinal region in children according to age groups.

DETAILED DESCRIPTION:
Regional anesthesia is frequently used in adults and children as part of multimodal analgesia or as a direct anesthesia method. Nowadays, these regional blocks can be applied more safely with the widespread use of ultrasound in daily clinical practice. Also, by identifying individual variations with ultrasound, the risk of block failure and possible complications has been minimized. Femoral nerve block and pericapsular nerve group block are now almost the first techniques used in hip and lower extremity surgeries or different indications. (1) Besides, these methods have become more advantageous in many aspects compared to spinal anesthesia in high-risk patients. However, to apply safe and successful regional anesthesia, both gross anatomy and sonoanatomy of the relevant region must be known well.

There are sufficient clinical and anatomical studies on these anesthesia methods applied in the inguinal region in adults, and there is no anatomical and anthropometric study in children. (2,3) However, well-known anatomic reference points for performing these blocks in adults may be different in children. (4) Therefore, with this study, we planned to develop appropriate anatomic reference points for these blocks in children by evaluating the relationship between sonography and inguinal region structures (such as distance, diameter measurement) in children's age groups.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients

Exclusion Criteria:

* a previous surgical history to the related area

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All pediatric patients within the predetermined age group
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
femoral artery and femoral nerve distance (mm) | 1 hour
  ultrasonographic measurements
Body weight (gr) | 1 hour
  measured at ward
height (cm) | 1 hour
  measured at ward

CONTACTS AND LOCATIONS:
Overall Officials: Hande Gurbuz, Assoc. Prof., Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Yıldırım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Result] Orozco S, Munoz D, Jaramillo S, Herrera AM. Pediatric use of Pericapsular Nerve Group (PENG) block for hip surgical procedures. J Clin Anesth. 2019 Nov;57:143-144. doi: 10.1016/j.jclinane.2019.04.010. Epub 2019 Apr 22. No abstract available. PMID 31022606
- [Result] Frkovic V, Warmlander SK, Petaros A, Spanjol-Pandelo I, Azman J. Finger width as a measure of femoral block puncture site: an ultrasonographic anatomical-anthropometric study. J Clin Anesth. 2015 Nov;27(7):553-7. doi: 10.1016/j.jclinane.2015.07.015. Epub 2015 Aug 31. PMID 26337562
- [Result] Vloka JD, Hadzic A, Drobnik L, Ernest A, Reiss W, Thys DM. Anatomical landmarks for femoral nerve block: a comparison of four needle insertion sites. Anesth Analg. 1999 Dec;89(6):1467-70. doi: 10.1097/00000539-199912000-00028. PMID 10589630
- [Result] Yoshimura M, Nakanishi T, Sakamoto S, Toriumi T. Age is a predictive factor in the femoral nerve positioning: an anatomical ultrasound study. J Anesth. 2018 Oct;32(5):777-780. doi: 10.1007/s00540-018-2544-2. Epub 2018 Aug 21. PMID 30132074
- [Derived] Gurbuz H, Colak T. Evaluation of inguinal sonoanatomy regarding pericapsular nerve group (PENG) block in children: the relation of femoral artery, femoral nerve, lateral femoral cutaneous nerve and iliopsoas notch. BMC Anesthesiol. 2025 Mar 31;25(1):144. doi: 10.1186/s12871-025-03020-2. PMID 40165082